CLINICAL TRIAL: NCT06601933
Title: Cognitive Training and Neuroplasticity in Mild Cognitive Impairment: COGIT-2 Trial
Acronym: COGIT-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Devangere P. Devanand, Professor of Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAU9623; 2R01AG052440-06A1 (NIH); WCG 20240282 (Other: Western-Copernicus Group (WCG) Institutional Review Board)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment (MCI); Cognitive Training
Keywords: Mild Cognitive Impairment; Cognitive Training; Crossword Puzzles; Health Education
MeSH Terms: conditions — Cognitive Dysfunction; Health Education | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Comparison of 3 treatment arms
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will know their treatment condition. Study investigators and clinicians and blinded research coordinator who administers outcomes assessments remain blind to treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): This sample will receive health education. The participant will read chapters from the book, "Living a Healthy Life with chronic conditions," 5th edition, by K Lorig, D Laurent, V Gonzalez, D Sobel, M Minor and M Gecht-Silver, and review chapters with the unblinded study coordinator.
  Interventions: Other: Cognitive Training
- Low Dose Crossword (Active Comparator): This sample will receive low dose crossword training with one crossword puzzle per week during the first 12 weeks on the Cognifit web-based platform. Subsequent booster sessions will occur at 20, 32, 42, 52, 64 and 78 weeks.
  Interventions: Other: Cognitive Training
- High Dose Crossword (Active Comparator): This sample will receive high dose crossword training. This sample will receive high dose crossword training with four crossword puzzles per week during the first 12 weeks on the Cognifit web-based platform, followed by booster sessions at 20, 32, 42, 52, 64 and 78 weeks.
  Interventions: Other: Cognitive Training

INTERVENTIONS:
Other: Cognitive Training — Participants (n=240) will be randomized to high dose crosswords, low dose crosswords, and health education at 1:1:1 ratio, stratified by site, age (< 70 and 70 years), and MCI status (early MCI and late MCI). In the two crossword puzzles conditions, after initial training to use the web-based platform, the participant will be assigned to do 12 weeks of crossword puzzles four times per week or 12 weeks of crossword puzzles once per week at home. After these 12 weeks, booster sessions will be either four or one 30-minute session(s) completed over 1 week. These booster sessions will occur at weeks 20, 32, 42, 52, 64, and 78. In-person assessments will occur at 0, 12, 32, 52, 78 weeks with one crossword puzzle session, which will count toward the booster session.
  Health education will involve reading chapters in a book on common illnesses and lifestyle, and a research staff member will review these chapters at the same assessment intervals as the crossword puzzles conditions.

SUMMARY:
Effective, clinically meaningful treatments are lacking for patients with mild cognitive impairment (MCI), which is associated with increased risk of transition to dementia. Cognitive training represents an important therapeutic strategy. In a previous study, crossword puzzles were found to be superior to computerized cognitive training on the primary cognitive outcome and function with decreased brain atrophy. Building on these findings, this study will evaluate and compare the impact of high dose crosswords (4 puzzles per week) to low dose crosswords (1 puzzle per week) and a health education control group on the cognition and function of participants.

DETAILED DESCRIPTION:
This study plans to enroll 240 participants with MCI: 75 at Columbia University, 60 at Duke, 60 at University of Miami, 45 at University of Washington. Participants will be randomized 1:1:1 to 4 crossword puzzles per week (high dose arm), 1 crossword puzzle per week (low dose arm), or health education (control arm). In the crossword groups, this initial intensive 12-week phase will be followed by booster sessions that will each comprise 30-minute sessions (1 or 4 sessions depending on assignment) completed over 1 week, and occur at weeks 20, 32, 42, 52, 64, and 78. In-person assessments will occur at 0, 12, 32, 52, 78 weeks. During weeks 0, 12, 32, 52, and 78, participants in the 4/week crosswords group will complete three sessions at home and the fourth in clinic, and participants in the 1/week group will complete one session in the clinic and none at home. During weeks 20, 42, and 64, participants will complete all sessions at home. The health education group will receive in-person sessions and assessments at weeks 0, 12, 32, 52, and 78 weeks, each for 30 min (same time frame as the crossword groups), and phone calls will be made, each for 30 min, at weeks 20, 42 and 64 to match the crossword groups (each 30 min). Unique features of the design: Evaluation of home-based crossword puzzles as the primary intervention; Comparison of two dose conditions to a comparison group; Health education comparison group with readings to mimic placebo in clinical trials; Stratification of random assignment by site, age, and early MCI/late MCI; Evaluation of MRI atrophy indices and plasma biomarkers of neurodegeneration (Neurofilament Light, Nfl) and Alzheimer Disease pathology (ptau-217).

ELIGIBILITY:
Inclusion Criteria:

1. Access to a home desktop or laptop computer or tablet at acceptable internet speed for the study duration.
2. Participants need to be 55 to 89 years of age (inclusive) at the time of informed consent.
3. Females need to be post-menopausal (last period more than 12 months earlier by history).
4. Subjective cognitive complaints, i.e., memory or other cognitive complaints, e.g., naming/language.
5. Meets criteria for cognitive impairment (CI), including either EMCI (early MCI) or LMCI (late MCI), defined as memory impairment documented by scoring below the education adjusted cutoff on the Logical Memory II subscale (Story A, Delayed Paragraph Recall) from the Wechsler Memory Scale - III (WMS-III) (the maximum score is 25). The criteria for MCI (includes EMCI and LMCI) and used in COGIT-2 are as follows: EMCI is defined by a WMS-III Logical memory delayed recall score of 3-6 with 0-7 years of education, score of 5-9 with 8-15 years of education, and score of 9-11 with 16 or more years of education. LMCI is defined by a WMS-III Logical Memory delayed recall score ≤ 2 with 0-7 years of education, score ≤ 4 with 8-15 years of education, and score ≤ 8 with ≥ 16 years of education.
6. Montreal Cognitive Assessment (MoCA) score ≥ 20/30.
7. An informant (relative, friend, other caregiver) who contacts the participant at least weekly is required to provide information about the participant's functioning. This can be a telephone informant in the case of participants who do not have a live-in informant or close significant other. If the informant drops out, an alternate informant can be designated by the participant but the new informant will need to sign the informant information sheet in person.
8. Must be English-speaking: Wide Range Achievement Test (WRAT3) score must indicate at least a 6th grade reading level with a score of ≥ 37.

Exclusion Criteria:

1. Diagnosis of dementia of any type.
2. Current clinical diagnosis of schizophrenia, schizoaffective disorder, psychosis, or bipolar I disorder (Diagnostic and Statistical Manual of Mental Disorders (DSM-5 TR) criteria).
3. Current unstable or untreated major depression, or active suicidality based on a Suicide Severity Rating Scale (C-SSRS Screen version: positive answer to question 1 or 2 followed by item 6 positive answer leads to exclusion. Negative answer to questions 1 and 2: interview ends and the participant is not excluded for active suicidality).
4. Current or recent (past 6 months) alcohol or substance use disorder (DSM-5 TR criteria).
5. Clinical stroke with residual neurological deficits. While we will not exclude participants with cerebrovascular disease or transient ischemic attacks (TIAs), we do not wish to include participants with a frank clinical stroke because it is not clear that this type of participant is similar to the MCI participant generally, and clear-cut neurological impairment, e.g., hemiplegia/hemiparesis or speech impairment, may compromise the ability to do the procedures and to complete the neuropsychological test battery.
6. Use of medications known to have a negative impact on cognition: benzodiazepines in lorazepam equivalents greater than or equal to 1 mg daily, narcotics, anticholinergics (ACB Calculator level 3 medication leads to exclusion), large number of sedating medications in combination. Medications with anticholinergic/antihistaminergic properties will be reviewed, e.g., low dose quetiapine (≤ 25 mg daily) will be permitted, but daily use of diphenhydramine or equivalent will be reviewed. Current use of lecanemab or donanemab will be exclusionary.
7. Presence of any of the following disorders: a) Central Nervous System Infections, with cerebrospinal fluid evidence of meningitis, encephalitis, or other infectious process; b) dementia of any type; c) Huntington's disease; d) Multiple sclerosis; e) Parkinson's disease; f) Other neurologic disorders with focal signs, e.g., amyotrophic lateral sclerosis.
8. Acute, severe unstable medical illness in the judgment of the clinician. For cancer, acutely ill participants (including those with metastases) are excluded, but history of successfully treated cancer does not result in exclusion.
9. Contraindication to MRI scan: MRI incompatible pacemakers and metal implants, any other contraindication to MRI. For participants with possible claustrophobia, they must be willing to do the MRI with adjunct lorazepam 0.5 mg to reduce anxiety. For participants who are recruited and are eligible for MRI but are unable to complete the baseline MRI, a repeat MRI for the same time-point can be attempted if the subject is willing. Baseline MRI is required for study inclusion.
10. Regular use of crosswords or formal computerized cognitive training platforms averaging once per week or more than once per week in the past year. Eligible participants who join the trial are instructed not to do these procedures on their own during the trial, i.e., independent of the study.
11. Participation concurrently in another therapeutic clinical trial of a cognitive enhancing drug or device or procedure.
12. Geriatric Depression Scale (Short Form) score of ≥ 6.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in ADASCog-14 (14-item Alzheimer's Disease Assessment Scale - Cognitive subscale) | Baseline, 78 weeks
  The ADASCog-14 is a brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia. It is one of the most widely used cognitive scales in clinical trials and is considered to be the "gold standard" for assessing antidementia treatments. The total score range is 0 to 90; a higher score indicates greater cognitive impairment.

SECONDARY OUTCOMES:
Change in Functional Activities Questionnaire (FAQ) score | Baseline, 78 weeks
  The FAQ is a patient-reported measure of cognitive impairment on difficulties in activities of daily living. The total score range is 0 to 30, with a higher score indicating greater impairment.
Change in MRI hippocampal volume | Baseline, 78 weeks
  The hippocampal volume is a measurement of brain atrophy. Hippocampal volume ranges from 0 to 10 cu cm with higher values indicating large hippocampal volume. Decrease in this measure indicates hippocampal atrophy.
Change in cortical thickness | Baseline, 78 weeks
  The cortical thickness is a measurement of brain atrophy. Values range from 0 to 1 with higher values indicating greater cortical thickness.

OTHER OUTCOMES:
Change in Preclinical Alzheimer Composite-5 (PACC5) | Baseline, 78 weeks
  PACC5 provides a comprehensive assessment of Alzheimer's disease-relevant cognitive impairment and to serve as a tool with validated sensitivity to detect cognitive decline over time. It is comprised of five tests: Mini-Mental State Examination (total score range 0-30), Wechsler Memory Scale-Revised Logical Memory Delayed Recall (total score range 0-25), Digit-Symbol Coding Test (total score range 0-93), Free and Cued Selective Reminding Test Free + Total Recall (total score range 0-96), and Category Fluency Test (graded by number of correct words belonging in the categories of animals, fruits, and vegetables; not graded on a scale). The PACC5 is computed as an averaged z-score of all five tests.
Change in Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale (ADCS-ADL-PI) | Baseline, 78 weeks
  The range of scores of the 15 items ADL question is 0-45 with higher scores indicating better performance. This is the outcome measure.
  In addition, there is a range of scores for the 5 items of physical function questions, which is 0-5 with higher scores indicating intact physical functioning.
plasma neurofilament light and ptau 217 | Baseline, 78 weeks
  Evaluate change in biomarkers over 78 weeks in the two crosswords groups and health education control group.
  Range = 0-999 ng/ml with higher values indicating more brain pathology.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for all measures will be shared among investigators in the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From October 15, 2024 until September 30, 2029

REFERENCES:
- [Background] Devanand DP, Goldberg TE, Qian M, Rushia SN, Sneed JR, Andrews HF, Nino I, Phillips J, Pence ST, Linares AR, Hellegers CA, Michael AM, Kerner NA, Petrella JR, Doraiswamy PM. Computerized Games versus Crosswords Training in Mild Cognitive Impairment. NEJM Evid. 2022 Dec;1(12):10.1056/evidoa2200121. doi: 10.1056/evidoa2200121. Epub 2022 Oct 27. PMID 37635843
- [Background] Motter JN, Pelton GH, D'Antonio K, Rushia SN, Pimontel MA, Petrella JR, Garcon E, Ciovacco MW, Sneed JR, Doraiswamy PM, Devanand DP. Clinical and radiological characteristics of early versus late mild cognitive impairment in patients with comorbid depressive disorder. Int J Geriatr Psychiatry. 2018 Dec;33(12):1604-1612. doi: 10.1002/gps.4955. Epub 2018 Jul 23. PMID 30035339
- [Background] Pfeffer RI, Kurosaki TT, Harrah CH Jr, Chance JM, Filos S. Measurement of functional activities in older adults in the community. J Gerontol. 1982 May;37(3):323-9. doi: 10.1093/geronj/37.3.323. PMID 7069156
- [Background] Liss JL, Seleri Assuncao S, Cummings J, Atri A, Geldmacher DS, Candela SF, Devanand DP, Fillit HM, Susman J, Mintzer J, Bittner T, Brunton SA, Kerwin DR, Jackson WC, Small GW, Grossberg GT, Clevenger CK, Cotter V, Stefanacci R, Wise-Brown A, Sabbagh MN. Practical recommendations for timely, accurate diagnosis of symptomatic Alzheimer's disease (MCI and dementia) in primary care: a review and synthesis. J Intern Med. 2021 Aug;290(2):310-334. doi: 10.1111/joim.13244. Epub 2021 Mar 31. PMID 33458891
- [Background] Segrave RA, Arnold S, Hoy K, Fitzgerald PB. Concurrent cognitive control training augments the antidepressant efficacy of tDCS: a pilot study. Brain Stimul. 2014 Mar-Apr;7(2):325-31. doi: 10.1016/j.brs.2013.12.008. Epub 2013 Dec 19. PMID 24486425
- [Background] Owens M, Koster EH, Derakshan N. Improving attention control in dysphoria through cognitive training: transfer effects on working memory capacity and filtering efficiency. Psychophysiology. 2013 Mar;50(3):297-307. doi: 10.1111/psyp.12010. Epub 2013 Jan 25. PMID 23350956
- [Background] Lohman MC, Rebok GW, Spira AP, Parisi JM, Gross AL, Kueider AM. Depressive symptoms and memory performance among older adults: results from the ACTIVE memory training intervention. J Aging Health. 2013 Dec;25(8 Suppl):209S-29S. doi: 10.1177/0898264312460573. Epub 2012 Sep 23. PMID 23006426
- [Background] Elgamal S, McKinnon MC, Ramakrishnan K, Joffe RT, MacQueen G. Successful computer-assisted cognitive remediation therapy in patients with unipolar depression: a proof of principle study. Psychol Med. 2007 Sep;37(9):1229-38. doi: 10.1017/S0033291707001110. Epub 2007 Jul 5. PMID 17610766
- [Background] Rozzini L, Costardi D, Chilovi BV, Franzoni S, Trabucchi M, Padovani A. Efficacy of cognitive rehabilitation in patients with mild cognitive impairment treated with cholinesterase inhibitors. Int J Geriatr Psychiatry. 2007 Apr;22(4):356-60. doi: 10.1002/gps.1681. PMID 17117398
- [Background] Harvey PD, Zayas-Bazan M, Tibirica L, Kallestrup P, Czaja SJ. Improvements in Cognitive Performance With Computerized Training in Older People With and Without Cognitive Impairment: Synergistic Effects of Skills-Focused and Cognitive-Focused Strategies. Am J Geriatr Psychiatry. 2022 Jun;30(6):717-726. doi: 10.1016/j.jagp.2021.11.008. Epub 2021 Nov 21. PMID 34924275
- [Background] Valenzuela MJ, Sachdev P. Brain reserve and dementia: a systematic review. Psychol Med. 2006 Apr;36(4):441-54. doi: 10.1017/S0033291705006264. Epub 2005 Oct 6. PMID 16207391
- [Background] Zissimopoulos J, Crimmins E, St Clair P. The Value of Delaying Alzheimer's Disease Onset. Forum Health Econ Policy. 2014 Nov;18(1):25-39. doi: 10.1515/fhep-2014-0013. Epub 2014 Nov 4. PMID 27134606
- [Background] Wolinsky FD, Jones MP, Dotson MM. Does Visual Speed of Processing Training Improve Health-Related Quality of Life in Assisted and Independent Living Communities?: A Randomized Controlled Trial. Innov Aging. 2020 Jul 31;4(4):igaa029. doi: 10.1093/geroni/igaa029. eCollection 2020. PMID 32964141
- [Background] Petersen RC. Mild cognitive impairment as a diagnostic entity. J Intern Med. 2004 Sep;256(3):183-94. doi: 10.1111/j.1365-2796.2004.01388.x. PMID 15324362
- [Derived] Wang LA, Goldberg TE, Harvey PD, Hanson AJ, Motter J, Andrews H, Qian M, Zhang R, Janis M, Doraiswamy PM, Devanand DP. Crossword puzzle training and neuroplasticity in mild cognitive impairment (COGIT-2): 78-week, multi-site, randomized controlled trial with cognitive, functional, imaging and biomarker outcomes. Int J Clin Trials. 2025 Apr-Jun;12(2):111-120. doi: 10.18203/2349-3259.ijct20251032. Epub 2025 Apr 11. PMID 40852373